CLINICAL TRIAL: NCT04108897
Title: Analysis of the Microbiome in Rosacea
Status: Active, not recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: IRB00210816
Record Dates: First submitted 2019-09-26; First posted 2019-09-30 (Actual); Last update posted 2025-06-13 (Actual); Status verified 2025-06

CONDITIONS: Rosacea
Keywords: rosacea; skin microbiome; gut microbiome; antimicrobial therapy
MeSH Terms: conditions — Rosacea | interventions — Doxycycline; Ivermectin

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (6):
- Doxycycline 40mg/day (Experimental): Doxycycline 40mg will be administered once a day per oral for 28 days.
  Interventions: Drug: Doxycycline
- Doxycycline 50mg/day (Experimental): Doxycycline 50mg will be administered once a day per oral for 28 days.
  Interventions: Drug: Doxycycline
- Doxycycline 100mg/day (Experimental): Doxycycline 100mg will be administered once a day per oral for 28 days.
  Interventions: Drug: Doxycycline
- Doxycycline 200mg/day (Experimental): Doxycycline 100mg will be administered twice a day per oral for 28 days.
  Interventions: Drug: Doxycycline
- Topical ivermectin(1%) (Experimental): Topical ivermectin will be applied once a day for 28 days.
  Interventions: Drug: Ivermectin Topical
- Control (No Intervention): No intervention will be performed.

INTERVENTIONS:
Drug: Doxycycline — The investigators will administer doxycycline to rosacea patients according to the dose of patients' assigned study arm.
  Arms: Doxycycline 100mg/day; Doxycycline 200mg/day; Doxycycline 40mg/day; Doxycycline 50mg/day
Drug: Ivermectin Topical — 1% topical ivermectin.
  Arms: Topical ivermectin(1%)

SUMMARY:
The skin and gut microbiome of rosacea patients differs from individuals without rosacea and that the microbiome suffers from unique derangements in rosacea patients following antibiotic therapy.

This study was proposed to examine microbial signatures of the skin and gut microbiome in patients with moderate to severe rosacea and to identify differences between microbe communities in patients with rosacea and volunteers without rosacea using 16S ribosomal ribonucleic acid (rRNA) polymerase chain reaction (PCR) amplification, sequencing and computational phylogenetics and to assess alterations in the gut and skin microbiota of patients with moderate to severe rosacea in response to varying formulations of antimicrobial treatment.

ELIGIBILITY:
Inclusion Criteria:

* Participants must be over the age of 18 years old.
* Participants must have a current diagnosis of moderate-to-severe erythematotelangiectatic or papulopustular rosacea or free of rosacea to serve as control.
* Participants must have the ability to understand and communicate with the investigator.
* Participants must be willing and comply with the requirements of the protocol.
* Participants must provide written informed consent

Exclusion Criteria:

* Subjects unable to provide informed consent.
* Subjects with significant medical history or concurrent illness that the investigator feels are not safe for study participation.
* Recently treated (4 weeks for topical antibiotics/steroids/other anti- inflammatory medications on the face, 8 weeks for systemic antibiotics/steroids/other immunosuppressive agents) or current (skin) diseases that would affect clinical evaluation and skin sampling.
* Subjects with a history of facial surgeries and cosmetic procedures (i.e. laser therapy, resurfacing, dermal fillers, and deep chemical peels) within 6 months.
* Subjects with facial features (i.e. significant hair growth) that would affect clinical evaluation and skin sampling.
* Participants with a history of chronic gastrointestinal disease, diabetes mellitus, cardiac disease or immunodeficiency disease.
* Intake of proton pump inhibitors, H2 receptor antagonists, laxatives, or antidiarrheal medication, NSAIDs, or antacids within 2 weeks prior to enrollment.
* Participants with a history of major surgery of the GI tract (5 years).
* Participants with a known hypersensitivity to tetracyclines or doxycycline or topical ivermectin
* Subjects unwilling to avoid facial washing for 24 hours prior to sampling and to come to sampling visit without make-up.
* Subjects with known allergy to lidocaine and epinephrine.
* Subjects with known bleeding disorders.
* Subjects with a history of keloids or excessive scarring.
* Pregnant subjects. Self-reporting will be used to determine whether a patient is pregnant

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2019-09-17 (Actual); Primary Completion 2027-09 (Estimated); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
Difference in skin and gut microbiome between rosacea and control | 2 months
  Differences between microbe communities in patients with rosacea and controls without rosacea will be assessed using a 16S rRNA PCR amplification, sequencing and computational phylogenetics.

SECONDARY OUTCOMES:
Change in skin and gut microbiome after 4-week of antimicrobial treatment in rosacea patients | Baseline, 28 days
  Alterations in the gut and skin microbiota of patients with rosacea in response to varying formulations of antimicrobial treatment will be assessed.

CONTACTS AND LOCATIONS:
Overall Officials: Anna Chien, Principal Investigator — Johns Hopkins University
Locations (1):
- Cutaneous Translational Research Program, Department of Dermatology, Baltimore, Maryland, United States